CLINICAL TRIAL: NCT01830543
Title: An Open-label, Randomized, Controlled, Multicenter Study Exploring Two Treatment Strategies of Rivaroxaban and a Dose-Adjusted Oral Vitamin K Antagonist Treatment Strategy in Subjects With Atrial Fibrillation Who Undergo Percutaneous Coronary Intervention
Brief Title: A Study Exploring Two Strategies of Rivaroxaban (JNJ39039039; BAY-59-7939) and One of Oral Vitamin K Antagonist in Patients With Atrial Fibrillation Who Undergo Percutaneous Coronary Intervention
Acronym: PIONEER AF-PCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100758; RIVAROXAFL3003 (Other: Janssen Scientific Affairs, LLC); 2012-001491-11 (EudraCT Number)
Record Dates: First submitted 2013-03-19; First posted 2013-04-12 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation; Percutaneous Coronary Intervention
Keywords: Atrial Fibrillation; Irregular heart beat; rivaroxaban; aspirin; clopidogrel; prasugrel; ticagrelor; vitamin K antagonist
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Rivaroxaban; Aspirin; acarboxyprothrombin; Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- rivaroxaban 2.5 mg twice daily (Experimental): rivaroxaban 2.5 mg tablet twice daily plus low-dose aspirin (ASA) 75 to 100 mg once daily and clopidogrel 75 mg tablet once daily (or prasugrel 10 mg tablet once daily or ticagrelor 90 mg tablet twice daily) followed by rivaroxaban 15 mg tablet (or 10 mg for subjects with moderate renal impairment) once daily plus low-dose ASA for 12 months
  Interventions: Drug: rivaroxaban 2.5 mg; Drug: rivaroxaban 15 mg; Drug: rivaroxaban 10 mg; Drug: aspirin (ASA); Drug: clopidogrel; Drug: prasugrel; Drug: ticagrelor
- vitamin K antagonist (VKA) (Experimental): dose-adjusted vitamin K antagonist (VKA) once daily (target International Normalized Ratio (INR) 2.0 to 3.0) plus low-dose ASA, 75 to 100 mg per day, and clopidogrel 75 mg once daily (or prasugrel 10 mg tablet once daily or ticagrelor 90 mg tablet twice daily) followed by dose-adjusted VKA once daily (target INR 2.0 to 3.0 or 2.0 to 2.5 at the investigator discretion) plus low-dose ASA for 12 months
  Interventions: Drug: aspirin (ASA); Drug: vitamin K antagonist (VKA); Drug: clopidogrel; Drug: prasugrel; Drug: ticagrelor
- rivaroxaban 15 mg once daily (Experimental): rivaroxaban 15 mg (or 10 mg for subjects with moderate renal impairment) once daily plus clopidogrel 75 mg tablet once daily (or prasugrel 10 mg tablet once daily or ticagrelor 90 mg tablet twice daily) for 12 months
  Interventions: Drug: rivaroxaban 15 mg; Drug: rivaroxaban 10 mg; Drug: clopidogrel; Drug: prasugrel; Drug: ticagrelor

INTERVENTIONS:
Drug: rivaroxaban 2.5 mg — One 2.5 mg tablet twice daily for up to twelve months
  Arms: rivaroxaban 2.5 mg twice daily
Drug: rivaroxaban 15 mg — One 15 mg tablet once daily for up to twelve months
  Arms: rivaroxaban 15 mg once daily; rivaroxaban 2.5 mg twice daily
Drug: rivaroxaban 10 mg — One 10 mg tablet once daily for up to twelve months
  Arms: rivaroxaban 15 mg once daily; rivaroxaban 2.5 mg twice daily
Drug: aspirin (ASA) — Low-dose aspirin tablet once daily for twelve months
  Arms: rivaroxaban 2.5 mg twice daily; vitamin K antagonist (VKA)
Drug: vitamin K antagonist (VKA) — Dose-adjusted VKA tablet (target International Normalized Ratio (INR) 2.0 to 3.0) once daily for twelve months
  Arms: vitamin K antagonist (VKA)
Drug: clopidogrel — One 75 mg tablet once daily for up to twelve months
Drug: prasugrel — One 10 mg tablet once daily for up to twelve months
Drug: ticagrelor — One 90 mg tablet twice daily for up to twelve months

SUMMARY:
The primary purpose of this study is to evaluate the safety for 2 different rivaroxaban treatment strategies and one Vitamin K Antagonist (VKA) treatment strategy utilizing various combinations of dual antiplatelet therapy (DAPT) or low-dose aspirin (ASA) or clopidogrel (or prasugrel or ticagrelor).

DETAILED DESCRIPTION:
This is an open-label (both physician and participant know the treatment that the participant receives), randomized (study medication is assigned by chance), multicenter clinical study assessing the safety of 2 rivaroxaban treatment strategies and one vitamin K antagonist (VKA) treatment strategy in participants, who have paroxysmal, persistent, or permanent non-valvular atrial fibrillation (AF) and have had a percutaneous coronary intervention (PCI) with stent placement.

A target of 2,100 participants will be randomized into the study, with approximately 700 participants in each treatment strategy group. The randomization will be stratified by the intended duration of DAPT (1, 6, or 12 months).

The study consists of a screening phase, a 12-month open-label treatment phase, and an end-of-treatment/early withdrawal visit. The total duration of participation in the study for each participant is approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented medical history of paroxysmal, persistent, or permanent non-valvular atrial fibrillation (AF)
* Have undergone percutaneous coronary intervention (PCI) procedure (with stent placement) for primary atherosclerotic disease
* Must have an international normalized ratio (INR) of 2.5 or below to be randomized
* Women must be postmenopausal before entry or practicing a highly effective method of birth control when heterosexually active
* Be willing and able to adhere to the prohibitions and restrictions specified in the study protocol

Exclusion Criteria:

* Have any condition that contraindicates anticoagulant or antiplatelet therapy or would have an unacceptable risk of bleeding, such as, but not limited to: platelet count <90,000/microliter at screening, history of intracranial hemorrhage, 12 month history of clinically significant gastrointestinal bleeding, non-VKA induced elevated prothrombin time (PT) at screening
* Have anemia of unknown cause with a hemoglobin level <10 g/dL (<6.21 mmol/L)
* Have a history of stroke or Transient Ischemic Attack (TIA)
* Have a calculated Creatinine Clearance (CrCl) <30 mL/min at screening
* Have known significant liver disease or liver function test (LFT) abnormalities
* Have any severe condition that would limit life expectancy to less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2124 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (348):
- United States (86):
  - Huntsville, Alabama
  - Los Alamitos, California
  - Mission Viejo, California
  - Oceanside, California
  - Riverside, California
  - Sacramento, California
  - San Francisco, California
  - Stockton, California
  - Thousand Oaks, California
  - Torrance, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Danbury, Connecticut
  - Washington D.C., District of Columbia
  - Atlantis, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Jacksonville, Florida
  - Port Charlotte, Florida
  - Safety Harbor, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Columbus, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Boise, Idaho
  - Hazel Crest, Illinois
  - Indianapolis, Indiana
  - Munster, Indiana
  - Hammond, Louisiana
  - Lake Charles, Louisiana
  - Slidell, Louisiana
  - Auburn, Maine
  - Bangor, Maine
  - Baltimore, Maryland
  - Detroit, Michigan
  - Lansing, Michigan
  - Mount Clemens, Michigan
  - Petoskey, Michigan
  - Ypsilanti, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Kalispell, Montana
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - Haddon Heights, New Jersey
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Ridgewood, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Peekskill, New York
  - Sanford, North Carolina
  - Bartlesville, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Portland, Oregon
  - Abington, Pennsylvania
  - Camp Hill, Pennsylvania
  - Doylestown, Pennsylvania
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sayre, Pennsylvania
  - York, Pennsylvania
  - Greenville, South Carolina
  - Mt. Pleasant, South Carolina
  - Rapid City, South Dakota
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Humble, Texas
  - Odessa, Texas
  - Plano, Texas
  - Layton, Utah
  - Charlottesville, Virginia
  - Manassas, Virginia
  - Midlothian, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Milwaukee, Wisconsin
  - Weston, Wisconsin
- Argentina (10):
  - Bahía Blanca
  - Buenos Aires
  - C.a.b.a.
  - Corrientes
  - Córdoba
  - La Plata
  - Resistencia
  - Rosario
  - Santa Fe
  - Vicente López
- Australia (7):
  - Chermside
  - Epping
  - Hobart
  - Kogarah
  - Liverpool
  - New Lambton
  - Wollongong
- Belgium (12):
  - Aalst
  - Bonheiden
  - Brasschaat
  - Bruges
  - Brussels
  - Genk
  - Ghent
  - Liège
  - Mechelen
  - Mol
  - Roeselare
  - Turnhout
- Brazil (14):
  - Belo Horizonte
  - Blumenau
  - Brasília
  - Campina Grande do Sul
  - Campinas
  - Curitiba
  - Marília
  - Passo Fundo
  - Porto Alegre
  - Recife
  - São José do Rio Preto
  - São Paulo
  - Uberlândia
  - Votuporanga
- Bulgaria (8):
  - Blagoevgrad
  - Burgas
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
  - Veliko Tarnovo
- Canada (15):
  - Edmonton, Alberta
  - Maple Ridge, British Columbia
  - New Westminster, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - St. John's, Newfoundland and Labrador
  - Greater Sudbury, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
  - Chicoutimi
  - Saint John
- Chile (5):
  - Alto
  - Concepción
  - Punta Arenas
  - Santiago
  - Temuco
- Czechia (12):
  - Brno
  - Hradec Králové
  - Jablonec Na Nisou
  - Karlovy Vary
  - Kladno
  - Litomyšl
  - Olomouc
  - Pilsen
  - Prague
  - Praha 10 N/A
  - Slaný
  - Uherské Hradiště
- Denmark (12):
  - Aalborg
  - Copenhagen
  - Esbjerg
  - Herlev
  - Herning
  - Hvidovre
  - Koege
  - Næstved
  - Odense
  - Roskilde
  - Svendborg
  - Vejle
- France (15):
  - Besancon Cedex Franche-Comté
  - Caen
  - Centrès
  - Chartres
  - Lille
  - Limoges
  - Marseille
  - Montfermeil
  - Nantes
  - Nîmes
  - Paris
  - Pau
  - Pessac
  - Poitiers
  - Toulouse
- Germany (16):
  - Bad Friedrichshall
  - Bad Nauheim
  - Berlin
  - Cologne
  - Dresden
  - Esslingen am Neckar
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Göttingen
  - Greifswald
  - Hamburg
  - Heidelberg
  - Limburg
  - Mannheim
  - Ulm
  - Witten
- Malaysia (4):
  - George Town
  - Johor Bahru
  - Kajang
  - Kuala Lumpur
- Mexico (9):
  - Aguascalientes
  - Guadalajara
  - León
  - México
  - Pachuca
  - Puebla City
  - Querétaro
  - Villahermosa
  - Zapopan
- Netherlands (12):
  - 's-Hertogenbosch
  - Alkmaar
  - Amsterdam
  - Amsterdam-Zuidoost
  - Breda
  - Delft
  - Gorinchem
  - Leiden
  - Maastricht
  - Nieuwegein
  - Sneek
  - Uden
- Poland (22):
  - Będzin
  - Bielsko-Biala
  - Chrzanów
  - Gdynia
  - Grodzisk Mazowiecki
  - Katowice
  - Krakow
  - Lodz
  - Mielec
  - Nowy Targ
  - Ostrowiec Świętokrzyski
  - Oświęcim
  - Płock
  - Rzeszow Poland
  - Starachowice
  - Starogard Gdański
  - Szczecin
  - Torun
  - Tychy
  - Ustroń
  - Warsaw
  - Zamość
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Târgu Mureş
  - Tg Mures
- Russia (16):
  - Arkhangelsk
  - Barnaul
  - Chita
  - Kemerovo
  - Krasnodar
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Perm
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Saratov
  - Syktyvkar
  - Tyumen
  - Yekaterinburg
- South Africa (4):
  - Cape Town
  - Centurion
  - Linksfield West, Johannesburg
  - Somerset West
- South Korea (9):
  - Busan
  - Daejeon
  - Gyeonggi-do
  - Incheon
  - Seongnam
  - Seoul
  - Suwon
  - Uijeongbu-si
  - Wŏnju
- Sweden (8):
  - Falun
  - Gothenburg
  - Jönköping
  - Lund
  - Malmo
  - Örebro
  - Stockholm
  - Umeå
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (9):
  - Ankara
  - Antalya
  - Bursa
  - Gaziantep
  - Istanbul
  - Istanbul Nap
  - Izmir
  - Kayseri
  - Sivas
- Ukraine (11):
  - Cherkassy
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Khemelnitskiy
  - Kyiv
  - Lviv
  - Odesa
  - Rivne
  - Uzhhorod
  - Zaporizhzhya
- United Kingdom (23):
  - Bath
  - Birmingham
  - Blackburn
  - Bradford
  - Clydebank
  - Cottingham
  - Coventry
  - Dorchester
  - Dundee
  - Edinburgh
  - Exeter
  - Hampshire
  - Harrow
  - High Wycombe
  - London
  - Middlesbrough
  - Norwich
  - Nottingham
  - Plymouth
  - Portsmouth
  - Torquay
  - Truro
  - Worcester

REFERENCES:
- [Derived] Kerneis M, Yee MK, Mehran R, Nafee T, Bode C, Halperin JL, Peterson ED, Verheugt FWA, Wildgoose P, van Eickels M, Lip GYH, Cohen M, Fox KAA, Gibson CM. Novel Oral Anticoagulant Based Versus Vitamin K Antagonist Based Double Therapy Among Stented Patients With Atrial Fibrillation: Insights From the PIONEER AF-PCI Trial. Circ Cardiovasc Interv. 2019 Nov;12(11):e008160. doi: 10.1161/CIRCINTERVENTIONS.119.008160. Epub 2019 Nov 11. PMID 31707805
- [Derived] Gibson WJ, Nafee T, Travis R, Yee M, Kerneis M, Ohman M, Gibson CM. Machine learning versus traditional risk stratification methods in acute coronary syndrome: a pooled randomized clinical trial analysis. J Thromb Thrombolysis. 2020 Jan;49(1):1-9. doi: 10.1007/s11239-019-01940-8. PMID 31535314
- [Derived] Kerneis M, Yee MK, Mehran R, Nafee T, Bode C, Halperin JL, Peterson ED, Verheugt FWA, Wildgoose P, van Eickels M, Lip GYH, Cohen M, Fox KAA, Gibson CM. Association of International Normalized Ratio Stability and Bleeding Outcomes Among Atrial Fibrillation Patients Undergoing Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2019 Feb;12(2):e007124. doi: 10.1161/CIRCINTERVENTIONS.118.007124. PMID 30704287
- [Derived] Chi G, Kerneis M, Kalayci A, Liu Y, Mehran R, Bode C, Halperin JL, Verheugt FWA, Wildgoose P, van Eickels M, Lip GYH, Cohen M, Peterson ED, Fox KAA, Gibson CM. Safety and efficacy of non-vitamin K oral anticoagulant for atrial fibrillation patients after percutaneous coronary intervention: A bivariate analysis of the PIONEER AF-PCI and RE-DUAL PCI trial. Am Heart J. 2018 Sep;203:17-24. doi: 10.1016/j.ahj.2018.06.003. Epub 2018 Jun 13. PMID 30015064
- [Derived] Chi G, Yee MK, Kalayci A, Kerneis M, AlKhalfan F, Mehran R, Bode C, Halperin JL, Verheugt FWA, Wildgoose P, van Eickels M, Lip GYH, Cohen M, Peterson ED, Fox KAA, Gibson CM. Total bleeding with rivaroxaban versus warfarin in patients with atrial fibrillation receiving antiplatelet therapy after percutaneous coronary intervention. J Thromb Thrombolysis. 2018 Oct;46(3):346-350. doi: 10.1007/s11239-018-1703-5. PMID 29943350
- [Derived] Kerneis M, Gibson CM, Chi G, Mehran R, AlKhalfan F, Talib U, Pahlavani S, Mir M, Bode C, Halperin JL, Nafee T, Peterson ED, Verheugt FWA, Wildgoose P, van Eickels M, Lip GYH, Fox KAA, Cohen M. Effect of Procedure and Coronary Lesion Characteristics on Clinical Outcomes Among Atrial Fibrillation Patients Undergoing Percutaneous Coronary Intervention: Insights From the PIONEER AF-PCI Trial. JACC Cardiovasc Interv. 2018 Apr 9;11(7):626-634. doi: 10.1016/j.jcin.2017.11.009. Epub 2018 Mar 14. PMID 29550085
- [Derived] Gibson CM, Mehran R, Bode C, Halperin J, Verheugt FW, Wildgoose P, Birmingham M, Ianus J, Burton P, van Eickels M, Korjian S, Daaboul Y, Lip GY, Cohen M, Husted S, Peterson ED, Fox KA. Prevention of Bleeding in Patients with Atrial Fibrillation Undergoing PCI. N Engl J Med. 2016 Dec 22;375(25):2423-2434. doi: 10.1056/NEJMoa1611594. Epub 2016 Nov 14. PMID 27959713
- [Derived] Gibson CM, Pinto DS, Chi G, Arbetter D, Yee M, Mehran R, Bode C, Halperin J, Verheugt FW, Wildgoose P, Burton P, van Eickels M, Korjian S, Daaboul Y, Jain P, Lip GY, Cohen M, Peterson ED, Fox KA. Recurrent Hospitalization Among Patients With Atrial Fibrillation Undergoing Intracoronary Stenting Treated With 2 Treatment Strategies of Rivaroxaban or a Dose-Adjusted Oral Vitamin K Antagonist Treatment Strategy. Circulation. 2017 Jan 24;135(4):323-333. doi: 10.1161/CIRCULATIONAHA.116.025783. Epub 2016 Nov 14. PMID 27881555
- [Derived] Gibson CM, Mehran R, Bode C, Halperin J, Verheugt F, Wildgoose P, van Eickels M, Lip GY, Cohen M, Husted S, Peterson E, Fox K. An open-label, randomized, controlled, multicenter study exploring two treatment strategies of rivaroxaban and a dose-adjusted oral vitamin K antagonist treatment strategy in subjects with atrial fibrillation who undergo percutaneous coronary intervention (PIONEER AF-PCI). Am Heart J. 2015 Apr;169(4):472-8.e5. doi: 10.1016/j.ahj.2014.12.006. Epub 2014 Dec 20. PMID 25819853

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivaroxaban 15 mg: Participants received rivaroxaban 15 milligram (mg) or 10 mg (for participants with moderate renal impairment [creatinine clearance (CrCl): 30 to less than (<) 50 milliliter per minute (mL/min)]) once daily plus background therapy with clopidogrel 75 mg once daily or alternate P2Y12 inhibitor (prasugrel 10 mg per day or ticagrelor 90 mg twice daily) for 12 months.
- Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD): Participants received rivaroxaban 2.5 mg twice daily plus background dual antiplatelet therapy (DAPT) with low-dose acetylsalicylic acid (ASA) 75 to 100 mg per day and clopidogrel 75 mg once daily (or alternate P2Y12 inhibitor [prasugrel or ticagrelor]) for an intended DAPT duration of 1, 6, or 12 months. Only participants with an intended DAPT duration of 1 or 6-month transitioned to receive rivaroxaban 15 mg or 10 mg (for participants with moderate renal impairment) once daily plus background single antiplatelet therapy with low-dose ASA for the rest of the period up to Month 12.
- Vitamin K Antagonist (VKA): Participants received dose adjusted (to a target of international normalized ratio [INR] 2.0 to 3.0 [or target INR 2.0 to 2.5]) vitamin K antagonist (VKA) [example warfarin, acenocoumarol; assigned by the investigator according to approved formulations) once daily plus background DAPT (clopidogrel 75 mg [or alternate P2Y12 inhibitor (prasugrel or ticagrelor)] plus low-dose ASA [75 to 100 mg] daily) for an intended DAPT duration of 1, 6, or 12 months. Only participants with an intended DAPT duration of 1 or 6-month transitioned to receive dose-adjusted VKA plus background single antiplatelet therapy with low-dose ASA for the rest of the period up to Month 12.
Period: Overall Study
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Started | 709 | 709 | 706
Treated | 696 | 706 | 697
Completed | 550 | 557 | 492
Not Completed | 159 | 152 | 214
Not completed — Subject Decision | 19 | 21 | 57
Not completed — Adverse Event | 91 | 77 | 76
Not completed — Death | 20 | 22 | 22
Not completed — Protocol Violation | 3 | 7 | 7
Not completed — Physician Decision | 11 | 5 | 12
Not completed — Withdrawal by consent | 3 | 3 | 3
Not completed — Other | 12 | 17 | 37

BASELINE CHARACTERISTICS:
Population: The intent-to-treat analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA) | Total
Number analyzed (Participants) | 709 | 709 | 706 | 2124
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (9.12) | 70 (9.11) | 69.9 (8.67) | 70.1 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 174 | 188 | 543
  Male | 528 | 535 | 518 | 1581
Region of Enrollment [Number; unit: participants]
  Argentina | 32 | 27 | 23 | 82
  Australia | 3 | 7 | 5 | 15
  Belgium | 14 | 18 | 20 | 52
  Brazil | 14 | 14 | 13 | 41
  Bulgaria | 67 | 80 | 74 | 221
  Canada | 23 | 24 | 19 | 66
  Chile | 5 | 7 | 6 | 18
  Czech Republic | 17 | 9 | 14 | 40
  Denmark | 2 | 2 | 8 | 12
  France | 33 | 26 | 25 | 84
  Germany | 96 | 98 | 101 | 295
  Italy | 26 | 26 | 20 | 72
  Korea, Republic of | 11 | 11 | 17 | 39
  Malaysia | 1 | 5 | 5 | 11
  Mexico | 7 | 3 | 3 | 13
  Netherlands | 24 | 17 | 27 | 68
  Poland | 71 | 78 | 69 | 218
  Romania | 15 | 16 | 19 | 50
  Russian Federation | 90 | 86 | 89 | 265
  Sweden | 15 | 14 | 18 | 47
  Taiwan, Province of China | 8 | 8 | 9 | 25
  Turkey | 11 | 14 | 18 | 43
  Ukraine | 19 | 24 | 17 | 60
  United Kingdom | 48 | 44 | 39 | 131
  United States | 56 | 49 | 46 | 151
  South Africa | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Significant Bleeding
Description: Clinically significant bleeding is a composite of Thrombolysis in Myocardial Infarction (TIMI) major bleeding, minor bleeding, and bleeding requiring medical attention (BRMA). TIMI major bleeding is defined as any symptomatic intracranial hemorrhage, clinically overt signs of hemorrhage (including imaging) associated with a drop in hemoglobin of greater than or equal to (>=) 5 grams per deciliter (g/dL) (or when the hemoglobin concentration is not available, an absolute drop in hematocrit of >=15 percent (%)). TIMI minor bleeding event is defined as any clinically overt sign of hemorrhage (including imaging) that is associated with a fall in hemoglobin concentration of 3 to less than (<) 5 g/dL (or, when hemoglobin concentration is not available, a fall in hematocrit of 9 percent to <15 percent). A BRMA event is defined as any bleeding event that requires medical treatment, surgical treatment, or laboratory evaluation, and does not meet criteria for a major or minor bleeding event.
Time Frame: Up to Month 12
Population: The safety analysis set is defined as all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 696 | 706 | 697
percentage of participants | 15.7 | 16.6 | 24.0
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.47 to 0.76]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.5 to 0.8]

2. Secondary Outcome: Percentage of Participants With Thrombolysis in Myocardial Infarction (TIMI) Major Bleeding
Description: TIMI major bleeding is defined as any symptomatic intracranial hemorrhage, Clinically overt signs of hemorrhage (including imaging) associated with a drop in hemoglobin of >= 5 g/dL (or when the hemoglobin concentration is not available, an absolute drop in hematocrit of >=15 percent).
Time Frame: Up to Month 12 and end of DAPT-Month 1, 6 and 12
Population: The safety analysis set is defined as all randomized participants who received at least 1 dose of study drug. Here, 'n' signifies number of participants analyzed at specific time-point in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 696 | 706 | 697
percentage of participants
  Up to Month 12 (n= 696, 706, 697) | 2.0 | 1.7 | 2.9
  End of DAPT-1 Month (n= 0, 108,113) | NA — Analysis at end of DAPT-1 month conducted only in participants who received DAPT as part of therapy. | 0.9 | 4.4
  End of DAPT-6 Month (n= 0, 248,243) | NA — Analysis at end of DAPT-6 month conducted only in participants who received DAPT as part of therapy. | 2.8 | 3.7
  End of DAPT-12 Month (n= 0, 350,341) | NA — Analysis at end of DAPT-12 month conducted only in participants who received DAPT as part of therapy. | 1.1 | 1.8
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.234, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.33 to 1.31]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.114, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.28 to 1.16]

3. Secondary Outcome: Percentage of Participants With Thrombolysis in Myocardial Infarction (TIMI) Minor Bleeding
Description: TIMI minor bleeding event is defined as any clinically overt sign of hemorrhage (including imaging) that is associated with a fall in hemoglobin concentration of 3 to <5 g/dL (or, when hemoglobin concentration is not available, a fall in hematocrit of 9 percent to <15 percent).
Time Frame: Up to Month 12 and end of DAPT-Month 1, 6 and 12
Population: The safety analysis set is defined as all randomized participants who received at least 1 dose of study drug. Here 'n' signifies number of participants analyzed at specific time-point in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 696 | 706 | 697
percentage of participants
  Up to Month 12 (n= 696, 706, 697) | 1.0 | 1.0 | 1.9
  End of DAPT-1 Month (n= 0, 108, 113) | NA — Analysis at end of DAPT-1 month conducted only in participants who received DAPT as part of therapy. | 0.9 | 1.8
  End of DAPT-6 Month (n= 0, 248, 243) | NA — Analysis at end of DAPT-6 month conducted only in participants who received DAPT as part of therapy. | 0.4 | 2.5
  End of DAPT-12 Month (n= 0, 350, 341) | NA — Analysis at end of DAPT-12 month conducted only in participants who received DAPT as part of therapy. | 1.4 | 1.5
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.144, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.2 to 1.28]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.134, Log Rank; Hazard Ratio (HR) = 0.5, 95% CI 2-sided [0.2 to 1.26]

4. Secondary Outcome: Percentage of Participants With Bleeding Requiring Medical Attention (BRMA)
Description: A BRMA event is defined as any bleeding event that requires medical treatment, surgical treatment, or laboratory evaluation, and does not meet criteria for a major or minor bleeding event.
Time Frame: Up to Month 12 and end of DAPT-Month 1, 6 and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 696 | 706 | 697
percentage of participants
  Up to Month 12 (n= 696, 706, 697) | 13.4 | 14.4 | 19.9
  End of DAPT-1 Month (n= 0, 108, 113) | NA — Analysis at end of DAPT-1 month conducted only in participants who received DAPT as part of therapy. | 16.7 | 18.6
  End of DAPT-6 Month (n= 0, 248, 243) | NA — Analysis at end of DAPT-6 month conducted only in participants who received DAPT as part of therapy. | 12.9 | 23
  End of DAPT-12 Month (n= 0, 350, 341) | NA — Analysis at end of DAPT-12 month conducted only in participants who received DAPT as part of therapy. | 14.9 | 18.2
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.47 to 0.8]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.002, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.52 to 0.86]

5. Secondary Outcome: Percentage of Participants With Composite of Adverse Cardiovascular Events (Cardiovascular Death, Myocardial Infarction (MI) and Stroke)
Description: Percentage of participants who experienced adverse cardiovascular events (cardiovascular death, myocardial Infarction (MI) and stroke) collectively, were assessed.
Time Frame: Up to Month 12 and end of DAPT-Month 1, 6 and 12
Population: The safety analysis set is defined as all randomized participants who received at least 1 dose of study drug. Here 'N' signifies number of participants who were evaluable for this outcome measure, 'n' signifies number of participants analyzed at specific time-point in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 694 | 704 | 695
percentage of participants
  Up to Month 12 (n= 694, 704, 695) | 5.9 | 5.1 | 5.2
  End of DAPT-1 Month (n= 0, 108, 112) | NA — Analysis at end of DAPT-1 month conducted only in participants who received DAPT as part of therapy. | 5.6 | 4.5
  End of DAPT-6 Month (n= 0, 248, 243) | NA — Analysis at end of DAPT-6 month conducted only in participants who received DAPT as part of therapy. | 6.5 | 3.7
  End of DAPT-12 Month (n= 0, 348, 340) | NA — Analysis at end of DAPT-12 month conducted only in participants who received DAPT as part of therapy. | 4 | 6.5
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.75, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.69 to 1.68]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.765, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.59 to 1.48]

6. Secondary Outcome: Percentage of Participants With Cardiovascular Death
Description: The percentage of participants with the first occurrence of cardiovascular death were evaluated.
Time Frame: Up to Month 12 and end of DAPT-Month 1, 6 and 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 694 | 704 | 695
percentage of participants
  Up to Month 12 (n= 694, 704, 695) | 2.2 | 2 | 1.6
  End of DAPT-1 Month (n= 0, 108, 112) | NA — Analysis at end of DAPT-1 month conducted only in participants who received DAPT as part of therapy. | 1.9 | 1.8
  End of DAPT-6 Month (n= 0, 248, 243) | NA — Analysis at end of DAPT-6 month conducted only in participants who received DAPT as part of therapy. | 2.4 | 1.6
  End of DAPT-12 Month (n= 0, 348, 340) | NA — Analysis at end of DAPT-12 month conducted only in participants who received DAPT as part of therapy. | 1.7 | 1.5
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.523, Log Rank; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.59 to 2.8]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.664, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.54 to 2.62]

7. Secondary Outcome: Percentage of Participants With Myocardial Infarction
Description: The percentage of participants with the first occurrence of Myocardial Infarction were evaluated.
Time Frame: Up to Month 12 and end of DAPT-Month 1, 6 and 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 694 | 704 | 695
percentage of participants
  Up to Month 12 (n= 694, 704, 695) | 2.7 | 2.4 | 3
  End of DAPT-1 Month (n= 0, 108, 112) | NA — Analysis at end of DAPT-1 month conducted only in participants who received DAPT as part of therapy. | 2.8 | 0.9
  End of DAPT-6 Month (n= 0, 248, 243) | NA — Analysis at end of DAPT-6 month conducted only in participants who received DAPT as part of therapy. | 2.8 | 2.5
  End of DAPT-12 Month (n= 0, 348, 340) | NA — Analysis at end of DAPT-12 month conducted only in participants who received DAPT as part of therapy. | 2 | 4.1
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.625, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.46 to 1.59]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.374, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.4 to 1.42]

8. Secondary Outcome: Percentage of Participants With Stroke
Description: The percentage of participants with the first occurrence of Stroke were evaluated.
Time Frame: Up to Month 12 and end of DAPT-Month 1, 6 and 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 694 | 704 | 695
percentage of participants
  Up to Month 12 (n= 694, 704, 695) | 1.2 | 1.4 | 1
  End of DAPT-1 Month (n= 0, 108, 112) | NA — Analysis at end of DAPT-1 month conducted only in participants who received DAPT as part of therapy. | 1.9 | 2.7
  End of DAPT-6 Month (n= 0, 248, 243) | NA — Analysis at end of DAPT-6 month conducted only in participants who received DAPT as part of therapy. | 2.4 | 0
  End of DAPT-12 Month (n= 0, 348, 340) | NA — Analysis at end of DAPT-12 month conducted only in participants who received DAPT as part of therapy. | 0.6 | 1.2
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.891, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.39 to 2.96]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.53, Log Rank; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.52 to 3.58]

9. Secondary Outcome: Percentage of Participants With Stent Thrombosis
Description: The percentage of participants with the first occurrence of stent thrombosis were evaluated.
Time Frame: Up to Month 12 and end of DAPT-Month 1, 6 and 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 694 | 704 | 695
percentage of participants
  Up to Month 12 (n= 694, 704, 695) | 0.7 | 0.9 | 0.6
  End of DAPT-1 Month (n= 0, 108, 112) | NA — Analysis at end of DAPT-1 month conducted only in participants who received DAPT as part of therapy. | 1.9 | 0.9
  End of DAPT-6 Month (n= 0, 248, 243) | NA — Analysis at end of DAPT-6 month conducted only in participants who received DAPT as part of therapy. | 1.6 | 0.4
  End of DAPT-12 Month (n= 0, 348, 340) | NA — Analysis at end of DAPT-12 month conducted only in participants who received DAPT as part of therapy. | 0 | 0.6
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.79, Log Rank; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.32 to 4.45]
Statistical Analysis 2: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) vs Vitamin K Antagonist (VKA); Test type: Superiority or Other; p = 0.574, Log Rank; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.4 to 5.09]

ADVERSE EVENTS:
Time Frame: Upto 12 months
Description: The Safety Analysis Set is defined as all randomized participants who received at least 1 dose of study drug.
Arm/Group | Rivaroxaban 15 mg | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) | Vitamin K Antagonist (VKA)
Serious Adverse Events (participants affected / at risk) | 237/696 | 225/706 | 271/697
Other Adverse Events (participants affected / at risk) | 174/696 | 210/706 | 234/697
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 15 mg (N=696) | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) (N=706) | Vitamin K Antagonist (VKA) (N=697)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 4
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypergammaglobulinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 3 | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 5 | 5 | 3
Angina Pectoris (Cardiac disorders) | 7 | 13 | 15
Angina Unstable (Cardiac disorders) | 16 | 12 | 23
Atrial Fibrillation (Cardiac disorders) | 13 | 21 | 23
Atrial Flutter (Cardiac disorders) | 0 | 5 | 4
Atrial Tachycardia (Cardiac disorders) | 0 | 2 | 1
Atrial Thrombosis (Cardiac disorders) | 4 | 1 | 0
Atrioventricular Block (Cardiac disorders) | 2 | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 1 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 2 | 2
Cardiac Disorder (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 21 | 16 | 31
Cardiac Failure Acute (Cardiac disorders) | 3 | 3 | 4
Cardiac Failure Chronic (Cardiac disorders) | 3 | 1 | 3
Cardiac Failure Congestive (Cardiac disorders) | 7 | 4 | 11
Cardiac Pseudoaneurysm (Cardiac disorders) | 0 | 1 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Cardiovascular Disorder (Cardiac disorders) | 2 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 3 | 5 | 2
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1 | 1
Coronary Artery Thrombosis (Cardiac disorders) | 0 | 1 | 0
Dressler's Syndrome (Cardiac disorders) | 0 | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 1 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 1 | 2
Palpitations (Cardiac disorders) | 0 | 1 | 2
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 2
Pericardial Haemorrhage (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 4 | 1 | 2
Supraventricular Tachycardia (Cardiac disorders) | 0 | 2 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Tachycardia Induced Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 2 | 1 | 1
Ventricular Tachycardia (Cardiac disorders) | 3 | 0 | 1
Deafness Neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Age-Related Macular Degeneration (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 3
Eye Haemorrhage (Eye disorders) | 0 | 1 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0
Acute Abdomen (Gastrointestinal disorders) | 0 | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 1 | 0 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Barrett's Oesophagus (Gastrointestinal disorders) | 0 | 0 | 1
Change of Bowel Habit (Gastrointestinal disorders) | 1 | 0 | 0
Colitis Microscopic (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Crohn's Disease (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastric Mucosa Erythema (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 3 | 3
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 2 | 1 | 1
Gastritis Erosive (Gastrointestinal disorders) | 0 | 2 | 2
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 1
Gastroduodenitis Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 7 | 7 | 9
Gastrointestinal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 3 | 0 | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 1 | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 4
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 1
Pancreatitis Chronic (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 4 | 2 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Tongue Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 1 | 2
Catheter Site Swelling (General disorders) | 1 | 0 | 0
Chest Discomfort (General disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 8 | 4 | 9
Death (General disorders) | 2 | 2 | 0
Device Failure (General disorders) | 1 | 0 | 0
Drug Intolerance (General disorders) | 1 | 0 | 0
Drug Resistance (General disorders) | 1 | 0 | 0
Drug Withdrawal Syndrome (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Gait Disturbance (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Medical Device Complication (General disorders) | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 3
Oedema Peripheral (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Sudden Cardiac Death (General disorders) | 1 | 1 | 0
Sudden Death (General disorders) | 2 | 1 | 3
Ulcer Haemorrhage (General disorders) | 0 | 0 | 1
Vascular Stent Occlusion (General disorders) | 0 | 0 | 1
Vascular Stent Restenosis (General disorders) | 0 | 1 | 1
Vascular Stent Thrombosis (General disorders) | 1 | 2 | 0
Vessel Puncture Site Haematoma (General disorders) | 1 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 2
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 1 | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 3
Hepatic Cyst (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis Acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic Shock (Immune system disorders) | 1 | 0 | 0
Abdominal Wall Abscess (Infections and infestations) | 2 | 0 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 2 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 3 | 1 | 1
Bronchitis Bacterial (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 2
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Encephalitis Viral (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0 | 0
Haematoma Infection (Infections and infestations) | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0 | 0
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Intervertebral Discitis (Infections and infestations) | 0 | 1 | 0
Liver Abscess (Infections and infestations) | 1 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 12 | 12 | 14
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2
Scrotal Abscess (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1
Septic Shock (Infections and infestations) | 1 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 3
Urosepsis (Infections and infestations) | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 5 | 6 | 7
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Pubis Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 2
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Biopsy Prostate (Investigations) | 0 | 0 | 1
Cardiac Stress Test (Investigations) | 0 | 1 | 0
Ejection Fraction Decreased (Investigations) | 0 | 1 | 0
Electrocardiogram Ambulatory Abnormal (Investigations) | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 2 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 4
Lipids Increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 0 | 1
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic Disorder (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatic Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adrenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gallbladder Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 2 | 4
Cerebral Infarction (Nervous system disorders) | 1 | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 4 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dizziness Postural (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0 | 1
Hemianopia (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Intercostal Neuralgia (Nervous system disorders) | 0 | 1 | 0
Intracranial Haematoma (Nervous system disorders) | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 5 | 2 | 4
Lacunar Infarction (Nervous system disorders) | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Parkinson's Disease (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 4 | 8
Tension Headache (Nervous system disorders) | 1 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 1 | 3
Viith Nerve Paralysis (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 2 | 1
Bladder Tamponade (Renal and urinary disorders) | 0 | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 1
Calculus Urethral (Renal and urinary disorders) | 0 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 3 | 4
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1
Prerenal Failure (Renal and urinary disorders) | 1 | 0 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 2 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0
Urethral Haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Urethral Stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 2 | 0
Cervical Polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 10
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Dyspnoea at Rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Angioplasty (Surgical and medical procedures) | 0 | 1 | 0
Aortic Valve Replacement (Surgical and medical procedures) | 0 | 0 | 1
Cardiac Ablation (Surgical and medical procedures) | 2 | 0 | 0
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 0 | 1 | 0
Cardiac Resynchronisation Therapy (Surgical and medical procedures) | 0 | 1 | 0
Cardioversion (Surgical and medical procedures) | 0 | 2 | 0
Cholecystectomy (Surgical and medical procedures) | 2 | 0 | 0
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 | 0 | 1
Coronary Artery Bypass (Surgical and medical procedures) | 1 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 0
Ileostomy Closure (Surgical and medical procedures) | 1 | 0 | 0
Implantable Defibrillator Insertion (Surgical and medical procedures) | 1 | 2 | 1
Knee Arthroplasty (Surgical and medical procedures) | 1 | 2 | 0
Mitral Valve Repair (Surgical and medical procedures) | 0 | 1 | 0
Percutaneous Coronary Intervention (Surgical and medical procedures) | 0 | 1 | 0
Renal Sympathetic Nerve Ablation (Surgical and medical procedures) | 1 | 0 | 0
Tooth Extraction (Surgical and medical procedures) | 1 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 1
Aortic Stenosis (Vascular disorders) | 1 | 1 | 0
Arterial Stenosis (Vascular disorders) | 0 | 2 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 1
Arteriovenous Fistula (Vascular disorders) | 0 | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Extremity Necrosis (Vascular disorders) | 0 | 1 | 0
Femoral Artery Occlusion (Vascular disorders) | 0 | 0 | 2
Haematoma (Vascular disorders) | 2 | 0 | 3
Haemorrhage (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 3 | 2 | 2
Hypertensive Crisis (Vascular disorders) | 1 | 3 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0
Intermittent Claudication (Vascular disorders) | 1 | 2 | 0
Lymphocele (Vascular disorders) | 1 | 0 | 0
Malignant Hypertension (Vascular disorders) | 0 | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 4 | 0 | 2
Peripheral Artery Thrombosis (Vascular disorders) | 2 | 0 | 0
Peripheral Embolism (Vascular disorders) | 0 | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 2 | 1
Peripheral Vascular Disorder (Vascular disorders) | 0 | 0 | 1
Shock Haemorrhagic (Vascular disorders) | 0 | 0 | 1
Venous Occlusion (Vascular disorders) | 1 | 0 | 0
Venous Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 15 mg (N=696) | Rivaroxaban 2.5 mg Twice Daily (BID)/15 mg Once Daily(QD) (N=706) | Vitamin K Antagonist (VKA) (N=697)
Angina Pectoris (Cardiac disorders) | 13 | 18 | 12
Diarrhoea (Gastrointestinal disorders) | 12 | 18 | 11
Gingival Bleeding (Gastrointestinal disorders) | 17 | 16 | 18
Oedema Peripheral (General disorders) | 14 | 12 | 18
Contusion (Injury, poisoning and procedural complications) | 13 | 35 | 25
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 2 | 10 | 14
Dizziness (Nervous system disorders) | 8 | 7 | 15
Haematuria (Renal and urinary disorders) | 18 | 14 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 21 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 67 | 59 | 82
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 16 | 15
Haematoma (Vascular disorders) | 21 | 31 | 61
Hypertension (Vascular disorders) | 17 | 2 | 7

LIMITATIONS AND CAVEATS:
First the stratification to either 1, 6 or 12 months of DAPT was based upon clinician choice and was not randomized. Secondly there was not sufficient power to definitively assess efficacy due to the modest number of adverse CV events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.